CLINICAL TRIAL: NCT05183516
Title: Evaluation of Tdap Vaccination and Plasma Biomarkers of Alzheimer's Disease
Brief Title: Tdap and Biomarkers of Alzheimer's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mindful Diagnostics and Therapeutics, LLC (Industry)
Collaborators: Infectious Disease Society of America (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tdap PANDA
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer Disease, Late Onset
Keywords: Tdap; Alzheimer's; biomarkers; B. pertussis; immune risk profile
MeSH Terms: conditions — Alzheimer Disease | interventions — Tetanus Toxoid

STUDY DESIGN:
Intervention Model Description: single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tdap (Experimental): Open label study, no placebo comparator
  Interventions: Biological: tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine

INTERVENTIONS:
Biological: tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine — Tdap is a combination vaccine that protects against three potentially life-threatening bacterial diseases: tetanus, diphtheria, and pertussis (whooping cough).
  Other Names: Tdap

SUMMARY:
Recently, the Tdap (tetanus toxoid, reduced diphtheria toxoid and acellular pertussis) vaccination was added to the list of immunizations associated with lower incidence of dementia. Plasma-based biomarkers for AD are a welcome alternative to expensive and invasive testing for Alzheimer's; these biomarkers include assessment of amyloid and tau and neurofilament light protein that assesses non-specific neurodegeneration. The investigators will test for these biomarkers, as well as some immune parameters, administer Tdap then repeat the blood tests in six months.

DETAILED DESCRIPTION:
A growing number of studies have consistently shown reduced incident risk of dementia associated with a variety of vaccinations. Most recently, data probes of medical claims from two large and disparate databases showed that vaccination for tetanus, diphtheria and pertussis (Tdap) was associated with a 42% decrease in dementia. Adult vaccination coverage remains low for most routinely recommended vaccines, including Tdap. This study will screen and qualify participants who do not meet the recommended frequency interval for Tdap vaccination. Participants will have consented to a review of their medical history (including vaccination history), a neurocognitive test and a battery of blood tests. Included in the blood testing will be plasma-based testing for amyloid, tau and neurofilament light protein. The study will be considered a pilot study; it will be an open-label trial. All participants will receive a single dose of the Tdap vaccine. Nine months after vaccination, participants will repeat the pre-vaccine blood tests. Primary objective will be the assessment of change in the Alzheimer's disease (AD) biomarkers. Bordetella pertussis (B. pertussis), the bacterium that causes whopping cough, is one of the targets of the Tdap vaccine. B. pertussis is a hypothesized infectious trigger of Alzheimer's disease (AD). A secondary objective of the study will be determination of present and past infection by B. pertussis via IgG testing as well as PCR of nasal swab and how this may relate to the Alzheimer biomarker responses to Tdap vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Immuno- competent
* Out of compliance for Tdap vaccine (none within 10 years).
* Ability of give informed consent.
* SAGE test 17 or greater

Exclusion Criteria:

* Immuno- compromised
* In compliance for Tdap vaccination (within 10 years).
* Known allergy to components of the Tdap vaccine.
* SAGE test <17

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Plasma Amyloid | start of study and 6 months
  Amyloid peptides 42/40 ratio
Change in Plasma Tau | start of study and 6 months
  a brain-specific protein that may be expected to leak from brain interstitial fluid to the plasma compartment in Alzheimer's disease as well as its preclincial and prodromal stages.

SECONDARY OUTCOMES:
Presence of B. pertussis | start of study and 6 months
  Nasal swab for the presence of B. pertussis
B. pertussis IgG | start of study
  Blood test for history of B. pertussis

CONTACTS AND LOCATIONS:
Overall Officials: Coad T Dow, MD, Principal Investigator — Mindful Diagnostics and Therapeutics
Locations (1):
- Mindful Diagnostics and Therapeutics, Eau Claire, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
No participant data will be shared with other researchers.

REFERENCES:
- [Background] Scherrer JF, Salas J, Wiemken TL, Jacobs C, Morley JE, Hoft DF. Lower Risk for Dementia Following Adult Tetanus, Diphtheria, and Pertussis (Tdap) Vaccination. J Gerontol A Biol Sci Med Sci. 2021 Jul 13;76(8):1436-1443. doi: 10.1093/gerona/glab115. PMID 33856020
- [Background] Rubin K, Glazer S. The pertussis hypothesis: Bordetella pertussis colonization in the pathogenesis of Alzheimer's disease. Immunobiology. 2017 Feb;222(2):228-240. doi: 10.1016/j.imbio.2016.09.017. Epub 2016 Sep 28. PMID 27692981
- [Background] Wiemken TL, Salas J, Morley JE, Hoft DF, Jacobs C, Scherrer JF. Comparison of rates of dementia among older adult recipients of two, one, or no vaccinations. J Am Geriatr Soc. 2022 Apr;70(4):1157-1168. doi: 10.1111/jgs.17606. Epub 2021 Dec 12. PMID 34897645
- [Result] West T, Kirmess KM, Meyer MR, Holubasch MS, Knapik SS, Hu Y, Contois JH, Jackson EN, Harpstrite SE, Bateman RJ, Holtzman DM, Verghese PB, Fogelman I, Braunstein JB, Yarasheski KE. A blood-based diagnostic test incorporating plasma Abeta42/40 ratio, ApoE proteotype, and age accurately identifies brain amyloid status: findings from a multi cohort validity analysis. Mol Neurodegener. 2021 May 1;16(1):30. doi: 10.1186/s13024-021-00451-6. PMID 33933117